CLINICAL TRIAL: NCT05595499
Title: A Phase II Randomized Double-Blind Placebo-Controlled Study of Fisetin to Improve Physical Function in Breast Cancer Survivors
Brief Title: Fisetin to Improve Physical Function in Stage I-III Breast Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-001170; NCI-2022-08061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016042 (NIH); R21CA277660 (NIH); K76AG074918 (NIH)
Record Dates: First submitted 2022-10-19; First posted 2022-10-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Specimen Handling; fisetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (fisetin) (Experimental): Patients receive fisetin PO on days 1, 2, and 3. Treatment repeats every 2 weeks for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Fisetin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (placebo) (Placebo Comparator): Patients receive placebo PO on the trial. on days 1, 2, and 3. Treatment repeats every 2 weeks for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Fisetin — Given PO
  Other Names: 3,3',4',7-Tetrahydroxyflavone; 7,3',4'-Flavon-3-ol
  Arms: Arm A (fisetin)
Drug: Placebo Administration — Given PO
  Arms: Arm B (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests whether fisetin works to improve physical function in women who have received chemotherapy for stage I-III breast cancer treatment. Fisetin is a naturally occurring substance that is found in strawberries and other foods. Fisetin eliminates cells that have undergone a process called senescence. Senescence is when a cell ages and permanently stops dividing but does not die. Over time, large numbers of these cells build up in tissues throughout the body and can release harmful substances that causes inflammation and damages nearby healthy cells. Studies have shown that chemotherapy causes a build-up of these senescent cells. Giving fisetin may eliminate senescent cells and improve physical function in postmenopausal women who have received chemotherapy for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of fisetin on physical function, as assessed using the 6-minute walk distance (6MWD), in frail older breast cancer survivors.

SECONDARY OBJECTIVES:

I. To determine the effect of fisetin on other measures of physical function (grip strength, short physical performance battery [SPPB], frailty phenotype, physical function component of the 36 item short form survey [SF-36]).

II. To determine the effect of fisetin on fatigability (Borg Rating of Perceived Exertion [RPE]).

III. To determine the effect of fisetin on neuropathy (Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 [QLQ-CIPN20]).

IV. To determine the effect of fisetin on cognitive function (Patient Reported Outcomes Measurement Information System [PROMIS] cognitive function short form).

V. To determine the effect of fisetin on health-related quality of life (SF-36).

VI. To determine the effect of fisetin on sleep (Insomnia Severity Index [ISI]).

VII. To determine the effect of fisetin on anxiety (GAD-7). VIII. To determine the effect of fisetin on depression (PHQ-8). IX. To determine the effect of fisetin on local and distant recurrence free survival.

X. To determine the effect of fisetin on breast cancer specific survival and overall survival.

XI. To evaluate the safety and tolerability of fisetin (physician and patient-reported Common Terminology Criteria for Adverse Events [CTCAEs]).

XII. To estimate rates of adherence to fisetin (pill diary).

EXPLORATORY OBJECTIVES:

I. To determine the effect of fisetin on p16 expression in peripheral CD3+ T-cells.

II. To determine the effect of fisetin on circulating senescence-associated secretory phenotype (SASP) inflammatory factors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive fisetin orally (PO) on days 1, 2, and 3. Treatment repeats every 2 weeks for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples throughout the trial.

ARM B: Patients receive placebo PO on the trial. on days 1, 2, and 3. Treatment repeats every 2 weeks for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up yearly for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Women who are postmenopausal at the start of study treatment.

Postmenopausal status will be established as follows:

* Women aged: >= 60 years OR
* Women aged < 60 years AND one of the following conditions is met:

  * They have not had any menstrual periods for at least 12 months in the absence of exogenous hormonal treatments, chemotherapy, and/or tamoxifen AND have serum estradiol and follicle-stimulating hormone (FSH) levels confirmed as being within the standard laboratory reference range for postmenopausal females.
  * They have documented irreversible bilateral oophorectomy.
  * They are receiving ovarian suppression with their breast cancer endocrine therapy

    * Women with a diagnosis of early-stage breast cancer (Stage I-III) treated with neo/adjuvant chemotherapy within 12 months of starting study treatment
    * No evidence of active/recurrent breast cancer or other serious chronic illnesses
    * Have evidence of frail health, defined as a diminished 6-minute walk distance (< 400m) at baseline
    * Platelets > 60,000/mm^3
    * White blood cell count > 2,000/mm^3
    * Absolute neutrophil count > 500/mm^3
    * Hemoglobin >= 8.0 g/dL
    * Total bilirubin =< 3.0 X upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) =< 4.0 x ULN
    * Alanine aminotransferase (ALT) =< 4.0 x ULN
    * Estimated glomerular filtration rate (eGFR) of >= 30mL/min/1.73m^2 per the Modification of Diet in Renal Disease (MDRD) calculation
    * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Cancer-directed chemotherapy, biological therapy, or immunotherapy within 30 days prior to the start of study treatment. Exceptions include: trastuzumab, pertuzumab, pembrolizumab, tamoxifen, ribociclib, abemaciclib, aromatase inhibitors and/or ovarian suppression.
* Surgery and/or radiation within the last 30 days of starting study treatment (Exception: invasive non- major procedures such as an outpatient biopsy)
* Subjects taking medications that are considered prohibited.

  * Exception: Subjects taking any of the medications listed in under "Temporary medication adjustment required" may participate if they are otherwise eligible AND the medication can be safely withheld (from immediately before the 1st study agent administration until at least 10 hours after the last study agent administration, for each dosing interval)
* On herbal and natural medications with possible senolytic properties (i.e., curcumin, kava kava, St. John's wort) and are unable or unwilling to hold its administration 2 days prior to and during study treatment dosing. Exceptions include cannabidiol (CBD), vitamins, probiotics, and fish oil. Other herbal and natural medications may be permitted or prohibited per clinician discretion
* Subjects taking potentially senolytic agents within the last year: fisetin, quercetin, luteolin, dasatinib or imatinib (or other tyrosine kinase inhibitors), piperlongumine, or navitoclax
* Subjects on therapeutic doses of anticoagulants (e.g., warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc.)
* Issues with tolerating oral medication (such as but not limited to, inability to swallow pills (g-tubes not allowed), malabsorption issues, ongoing nausea or vomiting during screening, history of Crohn's, gastric bypass/reduction, or celiac disease)
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Currently participating in another intervention research study seeking to improve functional status, alleviate frailty, muscle strength, exhaustion/fatigue, or cognitive function

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance (6MWD) | Baseline to day 60
  The 6MWD is a validated measure of physical function. Participants walk at their own pace for 6 minutes and distance (in meters) is measured at the end. Will be treated as a continuous variable. Its distribution will be transformed to normality as appropriate, Initially, a simple t-test will be used to compare the means of 6MWD at Day 60 by treatment groups.

SECONDARY OUTCOMES:
Change in grip strength | From baseline to day 60
  Generalized estimating equation (GEE) models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to access change in grip strength.
  Grip strength will be obtained using a hand dynamometer.
Change in Short Physical Performance Battery score | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to access change in short physical performance battery score.
Change in frailty phenotype | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in physical function component of 36-item Short Form (SF-36) | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in the Borg Rating of Perceived Exertion score | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy 20 scores | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in Patient Reported Outcomes Measurement Information System cognitive function short form score | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in composite SF-36 score | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in sleep (Insomnia Severity Index score) | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in anxiety (Generalized Anxiety Disorder-7 score) | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Change in depression (Patient Health Questionnaire-8 score) | From baseline to day 60
  GEE models will be fitted. The variables also will be dichotomized (e.g., < median, >= median) and GEE models for binary data used to test treatment effects over time.
Local recurrence free survival | Up to 3 years
  Will be compared between fisetin and placebo using the stratified log-rank test. The stratified Cox regression model will be used to obtain the estimate of the hazard ratio and the 95% confidence interval. The distributions of various survival endpoints will be estimated using the Kaplan-Meier method.
Distant recurrence free survival | Up to 3 years
  Will be compared between fisetin and placebo using the stratified log-rank test. The stratified Cox regression model will be used to obtain the estimate of the hazard ratio and the 95% confidence interval. The distributions of various survival endpoints will be estimated using the Kaplan-Meier method.
Breast cancer specific survival and overall survival | Up to 3 years
  Will be compared between fisetin and placebo using the stratified log-rank test. The stratified Cox regression model will be used to obtain the estimate of the hazard ratio and the 95% confidence interval. The distributions of various survival endpoints will be estimated using the Kaplan-Meier method.
Overall survival | Up to 3 years
  Will be compared between fisetin and placebo using the stratified log-rank test. The stratified Cox regression model will be used to obtain the estimate of the hazard ratio and the 95% confidence interval. The distributions of various survival endpoints will be estimated using the Kaplan-Meier method.
Adverse events rates | Up to 90 days
  Measured by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5. Adverse events will be determined at each time point per patient as the presence (yes/no) of toxicities (CTCAE v 5.0) of grade >= 2. The number of patients with adverse events will be compared by treatment arms using Fisher's exact test. GEE models for binary data will also be used to compare the proportion of patients with adverse events over time by treatment.
Adherence rate | From baseline up to 30 days
  Measured by pill diary. Treatment adherence (yes/no) for each patient at each time point will be determined. A patient will be considered adherent (coded 1) if she took all the required capsules within the allotted time, and non-adherent (coded 0) otherwise. The number of capsules taken in the allotted time out of the total required will also be recorded. Will then compare between treatments the proportion of adherent patients and the average proportion of capsules taken within the allotted time across patients at each time point using the t-test. Time point-specific analysis will be performed since conditions for pill-taking differ between the clinic (supervised) and patients' home (self-administered).

CONTACTS AND LOCATIONS:
Overall Officials: Mina S. Sedrak, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (7):
- United States (7):
  - UCLA Health Cancer Care in Alhambra, Alhambra, California
  - UCLA Health Beverly Hills Primary & Specialty Care, Beverly Hills, California
  - UCLA Health Burbank Primary & Specialty Care, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCLA Health Primary Care in Marina del Rey, Marina del Rey, California
  - UCLA Health Primary Care in Pasadena, Pasadena, California